CLINICAL TRIAL: NCT02297152
Title: A New Treatment for Premature Ejaculation? Case Series for a Desensitizing Masturbation Aid
Brief Title: A New Treatment for Premature Ejaculation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Sexológico Murciano (Other)
Responsible Party: Principal Investigator, Jesus Eugenio Rodríguez Martínez, Sexólogo, Instituto Sexológico Murciano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InstitutoSM
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Premature Ejaculation
Keywords: Premature ejaculation treatment; Sexual dysfunction; Intravaginal Ejaculatory Latency time; Masturbation aid; Ejaculatory disorders
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLIP HOLE (Other): The device Flip Hole is a masturbation aid made from Thermoplastic Elastomer (a silicone like substance) that the user inserts their penis in to for stimulation
  Interventions: Device: FLIP HOLE

INTERVENTIONS:
Device: FLIP HOLE — The subjects had to use the masturbator aid at least five times per week for six weeks, during a minimum of five minutes without never overcoming half daily hour and during intercourse. The device Flip Hole is a masturbation aid made from Thermoplastic Elastomer (a silicone like substance) that the user inserts their penis in to for stimulation.

SUMMARY:
The aim of study is to determine if they can produce increases in the IELT using a masturbator in subjects with premature ejaculation, producing improvements in the quality and satisfaction of the sexuality of the patient.

DETAILED DESCRIPTION:
From the assignment of the devices masturbation aid Flip Hole by the Japanese company TENGA® it was possible to begin to develop the study. To shape the patients sample was used to the active search of participants who met with the criteria of incorporation established for the participation in the study, from the publication of the study in different social media (Facebook, Twitter …) and the review of the database of the Instituto Sexológico Murciano patients' (ISM) who had represented previously with problems of premature ejaculation.

First interview with the participants was carried out where it informed them about the collaborative character in the study, together with the informed assent. To determine the suitability of the sample one administered ISM's Autobiographical questionnaire, the clinical Multiaxial Inventory of Millon-III (MCMI-III), and the Questionnaire of sexual satisfaction GRISS (Golombok Rust Sexual Inventory of Satisfaction), beside gathering a medical report of every patient to reject pathologies that they could interfere with the study.

Once established the number of participants, 15 males of ages included between 18 and 65 years, there was carried out a follow-up individualized for eight weeks from records of the IELT. During the first two weeks of research the subjects had to register the ejaculatory latency times during the manual masturbation and the intercourse being from the third week when they would use the device FLIP HOLE in the manual masturbation either alone or in company of the couple but never during the intercourse.

The subjects had to use the masturbator aid at least five times per week for six weeks, during a minimum of five minutes without never overcoming half daily hour and during intercourse. The device Flip Hole is a masturbation aid made from Thermoplastic Elastomer (a silicone like substance) that the user inserts their penis in to for stimulation.

The patients had to come weekly to ISM to deliver the weekly records and to be able to take a follow-up of the subjects along the process. Once finished eight weeks of the study one turned them to administer the questionnaire GRISS to evaluate if changes are produced in the sexual satisfaction of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets ISSM definition of PE
* Patient is 18 - 65 years

Exclusion Criteria:

* Patient has significant cardiovascular or neurological pathology.
* Patient has diabetes mellitus
* Patient is currently misusing alcohol/drugs
* Patient meets MCMI-III criteria for personality disorders and clinical syndromes

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the Intravaginal Ejaculatory Latency Time | 05/2014-09/2014 (during a minimum of five minutes without never overcoming half daily hour)
  During the first two weeks of research the subjects had to register the ejaculatory latency times during the manual masturbation and the intercourse being from the third week when they would use the device FLIP HOLE in the manual masturbation either alone or in company of the couple but never during the intercourse.
  The subjects had to use the masturbator aid at least five times per week for six weeks, during a minimum of five minutes without never overcoming half daily hour and during intercourse.

SECONDARY OUTCOMES:
Golombok Rust Sexual Inventory of Satisfaction | 05/2014-09/2014 (up to 4 months)
  subjects completing the questionnaire at the beginning of the investigation and when finalized using the Flip-Hole Masturbator device